CLINICAL TRIAL: NCT02720289
Title: Car Seat Education: What Works Best?
Brief Title: Video-Based Social Learning or Didactics for Car Seat Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 11-045
Record Dates: First submitted 2016-03-16; First posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Child Passenger Safety
Keywords: injury prevention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video-based social learning (Experimental): Video-based social learning class
  Interventions: Other: Video-based social learning class
- Traditional didactic (Active Comparator): Traditional didactic class
  Interventions: Other: Traditional didactic class

INTERVENTIONS:
Other: Video-based social learning class — Brief child passenger safety lecture by a child passenger safety technician and viewing of a car seat video.
  Arms: Video-based social learning
Other: Traditional didactic class — Child passenger safety lecture by a child passenger safety technician.
  Arms: Traditional didactic

SUMMARY:
This study compares a video-based social learning method to the traditional didactic method as a new way to teach caregivers about child passenger safety, including how to install a car seat. Half of the caregivers will attend the video-based social learning class, while the other half will attend the traditional didactic class. The investigators hypothesize that the video-based social learning method will lead to an equal or greater increase in caregiver child passenger safety proficiency when compared to the traditional didactic method.

DETAILED DESCRIPTION:
Previous studies have demonstrated the effectiveness of child passenger safety education, however, there is limited research identifying an optimal teaching method.

Social learning teaching methods are beneficial in promoting health-behavior change. The social learning theory hypothesizes that people learn and change their behavior by observation and modeling. The video used in the social learning method shows parents as role models methodically teaching proper car seat installation in a vehicle.

Traditionally, child passenger safety education classes are didactic in design, relying on lecture formats and live demonstrations. The didactic method includes verbal instructions from a child passenger safety technician about car seat installation.

ELIGIBILITY:
Inclusion Criteria:

* Parents or caregivers of car seat-age children (age zero to three years)
* Participation in the Kids Ride Safe Program

Exclusion Criteria:

* Spoke a language other than English or Spanish

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2011-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
5-Item Car Seat Installation Demonstration Measure | 30 minutes
  Each participant will install a car seat in their vehicle prior to, and immediately following, the intervention. A child passenger safety technician observing the installation and blinded to the intervention, will use this measure to evaluate the 5 areas of installation: direction, location, mechanism (seatbelt or lower anchors), harness position, and tether use. Participants will only be evaluated on installation demonstration areas relevant to their vehicle and car seat. Each item is scored correct or incorrect. Correct car seat installation is defined as all applicable items marked correct.

SECONDARY OUTCOMES:
5-Item Confidence in Car Seat Installation Ability Assessment | 30 minutes
  Self reported confidence in ability to correctly install a car seat with one question each for the 5 areas of installation: direction, location, mechanism (seatbelt or lower anchors), harness position, and tether use. Administered prior to, and immediately following, the intervention. The five question 10-point Likert scale assessment is scored 1-10 (1 = not confident; 10 = very confident). Confidence is defined as a 9 or 10 on the Likert scale.
15-Question Car Seat Installation Knowledge Test | 30 minutes
  Self reported objective knowledge test with questions about the four steps for child passenger safety (rear facing seat, forward facing seat, booster seat, and seat belt/shoulder harness) and the LATCH (Lower Anchors and Tethers for Children) system. The test contains true/false, multiple-choice, and fill in the blank questions. Each question is worth 1 point for a total of 15 points. Adequate car seat knowledge is defined as 10 or more questions correct.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Kuroiwa, MHI, Principal Investigator — Phoenix Children's Hospital
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States